CLINICAL TRIAL: NCT00495820
Title: Methylphenidate for Apathy in Alzheimer's Dementia: A Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBB-011-06F
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Alzheimer's Disease; Apathy; Dementia
Keywords: Alzheimer's Disease; Apathy; Dementia; Methylphenidate
MeSH Terms: conditions — Alzheimer Disease; Lethargy; Dementia | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Methylphenidate
  Interventions: Drug: Methylphenidate
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Subject will receive 5mg twice a day for two weeks then 10mg twice a day until week 12 of the study.
  Other Names: Ritalin
  Arms: Arm 1
Other: Placebo — Standard inactive pill.
  Arms: Arm 2

SUMMARY:
The purpose of the study is to determine the efficacy of methylphenidate over placebo in treating apathy in patients with Alzheimer's dementia. Apathy is one of the earliest and most profound disturbances that occur in Alzheimer's dementia (AD).

Hypotheses: 1. Methylphenidate (MPH) will improve apathy significantly more than placebo in AD.

2. Successful treatment of apathy will improve Instrumental Activities of Daily Living (IADLs), and caregiver burden.

DETAILED DESCRIPTION:
Objective: Apathy is one of the earliest and most profound disturbances that occur in Alzheimer's dementia (AD). Based on promising preliminary data from our open-label pilot study we propose a double blind, placebo-controlled randomized clinical trial of methylphenidate for treatment of apathy in AD.

Research Design: Randomized double blind, placebo-controlled study which will evaluate the effect of methylphenidate on apathy and also the impact of improvement of apathy on caregiver burden and functional status.

Hypotheses: 1. Methylphenidate will improve apathy significantly more than placebo in AD.

2. Successful treatment of apathy will improve Instrumental Activities of Daily Living (IADLs), and caregiver burden.

Methodology: 60 patients with apathy in the context of AD will be recruited over the next three years. In our proposed study patients will be recruited from relevant clinics at the Omaha Veterans Affairs Medical Center (VAMC) including clinics in Geriatric Psychiatry, Neurology, Primary Care and Geriatric Medicine. 30 patients each with AD and apathy will be randomly assigned to placebo or MPH. All patients in the methylphenidate arm will be started at 5mg twice daily and titrated to 10mg twice daily at two weeks. Patients will be continued in this arm for 12 weeks followed by a 2-week discontinuation phase. Patients will be assessed on regular intervals using the Apathy Evaluation Scale, Instrumental Activities of Daily Living, Zarit Burden Scale and Mini Mental State Examination.

Findings: None, the study is not complete.

Clinical Relationships: While memory is the key cognitive problem in AD, apathy is the key behavioral problem. Apathy is characterized by indifference, disengagement, passivity, and lack of enthusiasm, interest, empathy and interpersonal involvement. Apathy is the most common, one of the earliest and probably the most persistent of behavioral problems in AD. Apathy is the most disturbing behavior to caregivers and has the greatest impact on functional status and caregiver burden.

Despite this, apathy as a behavioral problem has largely been neglected. Most of the research directed towards behavioral problems in dementia is targeted towards more visible behaviors such as agitation, and psychosis. Remarkably, there are no published randomized, double blind, placebo controlled studies in the treatment of apathy associated with AD.

Impact/Significance: Around 1.4 million veterans suffer from apathy in association with AD. Apathy is a strong predictor for functional decline and caregiver burden. Treatment of apathy is remarkably understudied and is absolutely critical to allow veterans to maximize their functional status, social engagement and quality of life, and thus delaying placement in assisted living or nursing home settings.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of dementia of the Alzheimer type (DSM-IV Text Revision (TR) criteria)
2. Mini-mental state examination (MMSE) >18, but <29
3. Apathy Evaluation Scale (AES) score of more than 40
4. Ability to provide informed consent by either the patient or caregiver.
5. If subjects are being treated with antidepressants, they should be on a stable dose of antidepressants for at least two months prior to the enrollment into the study.
6. If subjects are being treated with cholinesterase inhibitors and memantine, they should be on stable dose of those medications at least four months prior to the enrollment into the study.

Exclusion Criteria:

1. Patient currently taking methylphenidate or hypersensitivity or prior significant adverse events with methylphenidate.
2. Patients currently taking Adderall (amphetamine mixed salts) or Dexedrine (dextroamphetamine sulphate) or any other amphetamine product.
3. Uncontrolled hypertension (BP > 140/90) or tachycardia (100) at screening visit
4. Patients with frontotemporal dementia
5. Patients meeting criteria for Major Depressive Disorder on the Mini International Neuropsychiatric Inventory (MINI)
6. Patients with active psychosis as determined by MINI
7. Patients currently being treated with antipsychotics
8. History of uncontrolled seizure disorder
9. History of malignant hypertension, symptomatic cardiovascular disease, cardiomyopathy, known structural cardiac defect or medically unstable arrhythmias.
10. History of Tourette's syndrome or presence of motor tics
11. Patients with glaucoma
12. Patients taking monoamine oxidase inhibitors (MAOIs)
13. Patient taking clonidine

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prasad R. Padala, Principal Investigator — VA Medical Center, Omaha
Locations (1):
- VA Medical Center, Omaha, Omaha, Nebraska, United States

REFERENCES:
- [Result] Padala PR, Burke WJ, Shostrom VK, Bhatia SC, Wengel SP, Potter JF, Petty F. Methylphenidate for apathy and functional status in dementia of the Alzheimer type. Am J Geriatr Psychiatry. 2010 Apr;18(4):371-4. doi: 10.1097/JGP.0b013e3181cabcf6. PMID 20220576
- [Derived] Padala PR, Padala KP, Lensing SY, Ramirez D, Monga V, Bopp MM, Roberson PK, Dennis RA, Petty F, Sullivan DH, Burke WJ. Methylphenidate for Apathy in Community-Dwelling Older Veterans With Mild Alzheimer's Disease: A Double-Blind, Randomized, Placebo-Controlled Trial. Am J Psychiatry. 2018 Feb 1;175(2):159-168. doi: 10.1176/appi.ajp.2017.17030316. Epub 2017 Sep 15. PMID 28945120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 subjects meeting the inclusion and exclusion criteria were recruited from outpatient clinics at the Nebraska Western Iowa Health Care System between 2006-2009.
Groups:
- Arm 1: Methylphenidate
  Methylphenidate: Subject will receive 5mg BID for two weeks then 10mg BID until week 12 of the study.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.5 (7.9) | 76.1 (8.4) | 76.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Apathy Evaluation Scale [Mean (Standard Deviation); unit: units on a scale] — Range: 18-72 Higher scores indicate worse apathy
  units on a scale | 51.9 (7.1) | 47.6 (5.8) | 49.7 (6.8)
Mini-mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Range 0-30. Higher scores indicate better cognition
  units on a scale | 23.7 (2.5) | 24 (2.6) | 23.8 (2.5)
Modified Mini-Mental State Examination (3MS) [Mean (Standard Deviation); unit: units on a scale] — Range 0-100. Higher scores indicate better cognition
  units on a scale | 80.1 (9) | 82.6 (10) | 81.3 (9.5)
Activities of Daily Living [Mean (Standard Deviation); unit: units on a scale] — Range 0-24. Higher scores indicate better independence in performing activities of daily living.
  units on a scale | 21.3 (2.7) | 22.9 (2.2) | 22 (2.6)
The Executive Interview (EXIT-25) [Mean (Standard Deviation); unit: units on a scale] — Range: 0-50, higher scores indicate worsening of executive function.
  units on a scale | 16.9 (6.3) | 16.8 (6.6) | 16.8 (6.4)
Zarit Burden Scale [Mean (Standard Deviation); unit: units on a scale] — Range 0-88. Higher scores indicate higher caregiver burden.
  units on a scale | 28.1 (13) | 25.3 (13.3) | 26.9 (13)
Clinical Global Impression-severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — Range 0-7, higher scores indicating worsening of condition.
  units on a scale | 5.5 (0.6) | 5.1 (0.6) | 5.3 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Apathy Evaluation Scale Score at 12 Weeks
Description: The Apathy Evaluation Scale (AES) has been specifically developed to assess apathy and discriminate it from depression. This 18 item scale with score ranging from 18 to 72, assesses apathy in behavioral, cognitive and emotional domains over the previous four weeks. Higher scores indicate worsening apathy.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Methylphenidate Group: Subjects randomized to this group received methylphenidate
- Placebo Group: Subjects randomized to this group received placebo
Arm/Group | Methylphenidate Group | Placebo Group
Number analyzed (Participants) | 30 | 30
units on a scale | 38.2 (9.1) | 43.6 (7.5)
Statistical Analysis 1: Comparison: Methylphenidate Group vs Placebo Group; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Mini-mental State Examination (MMSE) at 12 Weeks
Description: Mini-mental State Examination (MMSE) is a commonly used screening measure for cognition with questions pertaining to orientation, registration, recall, visuo-spatial construction, attention span etc. Score on MMSE ranges from 0-30, higher scores indicating improving cognition
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Group | Placebo Group
Number analyzed (Participants) | 30 | 30
units on a scale | 25.8 (2.7) | 23.6 (4)
Statistical Analysis 1: Comparison: Methylphenidate Group vs Placebo Group; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

3. Secondary Outcome: Clinical Global Impression
Description: The Clinical Global Impression scale is an observational scale of global evaluation, which assesses the change in degree of illness in relation to the original assessment. The severity sub-scale reported below ranges from 1-7 wherein higher scores indicate worsening severity of illness.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate Group | Placebo Group
Number analyzed (Participants) | 30 | 30
units on a scale | 3.9 (1.1) | 4.8 (0.6)

ADVERSE EVENTS:
Groups:
- Placebo Group: Subjects randomized to this group received methylphenidate
Arm/Group | Methylphenidate Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 14/30 | 16/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate Group (N=30) | Placebo Group (N=30)
Nausea (Gastrointestinal disorders) | 5 (7) | 4 (4)
Increased blood pressure (Cardiac disorders) | 2 (3) | 1 (1)
Weight loss (Gastrointestinal disorders) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 3 (3) | 5 (6)
restlessness (Nervous system disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (3)

LIMITATIONS AND CAVEATS:
Small sample size and short duration of the study are two important limitations of the study. All male subjects in the study also make it difficult to generalize the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes